CLINICAL TRIAL: NCT05335850
Title: Meditation and Breathing for Mental Health in Parkinson's Disease Patient
Brief Title: Yoga for Mental Health in Parkinson's Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Balachundhar Subramaniam, Professor of Anesthesia, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2022P000212
Record Dates: First submitted 2022-04-06; First posted 2022-04-19 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Stress; Anxiety; Depression; Parkinson Disease
Keywords: Stress; Anxiety; Depression; Parkinson's Disease; Meditation; Breathing; Isha Kriya; Yoga; Mental Health
MeSH Terms: conditions — Anxiety Disorders; Depression; Parkinson Disease; Respiratory Aspiration; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: Crossover Assignment A partial crossover model ensures that both experimental and waitlisted control group participants get to experience the effects of a proposed intervention. For our study, we are providing these practices as an intervention and both experimental and waitlisted control group participants get to experience the benefits of meditation and breathing exercises.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Breathing and Wellness Webinar: a Yogic Breathing practice (Nadi Shuddhi) and two guided meditations (Isha Kriya and Nada Yoga).
  Interventions: Behavioral: Isha Kriya; Behavioral: Nadi Shuddhi; Behavioral: Nada Yoga
- Waitlisted Control Group (Active Comparator): This group will be asked to wait for 6 weeks before being introduced to the Breathing and Wellness Webinar intervention which includes a Yogic Breathing practice (Nadi Shuddhi) and two guided meditations (Isha Kriya and Nada Yoga).
  Interventions: Other: Routine Daily Activity

INTERVENTIONS:
Behavioral: Isha Kriya — Isha Kriya is a 15-minute guided meditation that incorporates the breath and the awareness to create mental clarity and health, to be practiced at least once (ideally twice) daily.
  Arms: Intervention Group
Behavioral: Nadi Shuddhi — Nadi Shuddhi is a gentle 4-minute breathing practice for creating mental balance and relaxation, to be practiced for a minimum of 4 minutes daily.
  Arms: Intervention Group
Behavioral: Nada Yoga — Nada Yoga is a 6-minute meditation that uses sound to create balance and stability in the body and mind.
  Arms: Intervention Group
Other: Routine Daily Activity — Participants in the control group are asked to perform routine daily activities until enrolled into the intervention arm.
  Participants in the control group are asked to perform routine daily activities until enrolled into the intervention arm.
  Arms: Waitlisted Control Group

SUMMARY:
This study is a waitlisted randomized controlled trial. We aim to assess the level of compliance for those learning the intervention and to evaluate the impact of the practice on neuropsychological and somatic outcomes using validated scales. Enrollment into the study will be ongoing until we are able to get a sufficient sample size as described in the "Statistical Consideration" section. Upon enrollment and randomization, surveys will be administered to both the intervention and control groups at four time-points: baseline, T2, T3, and T4, each of which are 6 weeks apart. Compliance data will be collected weekly for 12 weeks for both groups.

DETAILED DESCRIPTION:
Mental health issues caused by emotional and behavioral changes are common among people diagnosed with Parkinson's disease. Research from the Parkinson's Foundation's Parkinson's Outcomes Project has found that anxiety and depression play a key role in the disease's impact on people's quality of life. The death of dopamine-producing cells in the brain affects both movement and mood. As a result, both anxiety and depression are common non-motor symptoms of the disease rather than reactions to the diagnosis.

According to the Parkinson's Outcomes Project, during their illness:

* At least 50% of people will experience some form of depression
* At least 40% of people will experience an anxiety disorder

Forms of anxiety include Generalized Anxiety Disorder, Anxiety Attacks, Social Avoidance, and OCD1. Depression in Parkinson's disease often manifests as dissatisfaction with life, sadness, irritability, pessimism, and suicidal thoughts.

Meditative techniques have been shown to effectively reduce symptoms of anxiety and depression. Treating these non-motor symptoms can have a positive impact on people with Parkinson's disease by decreasing disability and improving their quality of life.

The purpose of this study is to investigate the impact of a set of simple, safe and scalable, digitally delivered meditation and breathing practices on the neuropsychological and movement disorder symptoms in patients with Parkinson's Disease over a period of 18-20 weeks. The intervention consists of a Yogic Breathing practice (Nadi Shuddhi) and two guided meditations (Isha Kriya and Nada Yoga). Our recent studies using similar interventions have shown feasibility and acceptance as well as Improved perceived stress in healthy subjects.

The subjects will be randomized into two groups after they agree to participate in the study, an intervention group (Group 1) and a waitlisted control group (Group 2). Both groups will learn and practice the intervention for 12 weeks total.The intervention is made of a Yogic Breathing practice (Nadi Shuddhi) and two guided meditations (Isha Kriya and Nada Yoga). Both groups will also take study surveys at 4 timepoints which are each 6 weeks apart (Baseline, T2, T3, and T4). The study surveys consist of an online survey and a clinician, phone administered survey.

This trial will be conducted in 2 phases:

Phase 1: If participants are in the intervention group, they will be asked to learn the practices first for 6 weeks, from T1-T2. They will be asked to complete weekly activity logs for these 6 weeks and the study survey at T2 (6 weeks after learning the intervention). Participants in the waitlisted control group will be asked to perform their regular daily routine as they wait to be enrolled into the intervention at T2 (6 weeks after Baseline). The waitlisted control group will also complete the study survey at T2.

Phase 2: After T2, the intervention group is no longer asked to attend weekly review webinars but they will continue to do weekly activity logs for 6 weeks until until T3. They will then complete the study survey at T3. After T3, they will not be sent any activity logs for the next 6 weeks until T4. At T4, they will be asked to complete the study survey and satisfaction survey. The waitlisted control group will begin the intervention at T2 and will attend review webinars for 6 weeks until T3 at which they will complete the study survey. After T3, they are no longer asked to attend weekly webinars but they will continue to do weekly activity logs for 6 weeks until until T4. At T4, they will be asked to complete the study survey and satisfaction survey.

ELIGIBILITY:
Inclusion Criteria:

* Age above 18
* Interested in attending the Breath, Sound, and Meditation Webinar
* Diagnosed with Parkinson's Disease
* PAS score of 12 or higher
* Able to read and comprehend English.
* Physically and mentally able to participate in the study procedure
* Currently residing in the United States.

Exclusion Criteria:

* Severe stage of PD
* Any medically limiting diagnosis that prevents a patient from doing the intervention or completing the assessments as determined by the PI such as severe Major Depression (under medication), Schizophrenia, Bipolar disorder.
* Not able to self-consent to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2022-10-18 (Actual); Primary Completion 2024-09-12 (Actual); Study Completion 2024-09-25 (Actual)

PRIMARY OUTCOMES:
Change in Compliance | For Phase 1 analysis: Baseline to week 6. For Phase 2 analysis: Baseline to week 18.
  The weekly compliance questionnaire is a tool which helps the participants to keep track of their activities each week. This enables the study team to measure compliance and protocol adherence by the participants by collecting information on their routine activity practiced and its frequency. This will be reported in "Number of days an intervention was practiced in a week". Participants completing at least 4 days of activity would be considered as compliant for that week.
Change in Anxiety | For Phase 1 analysis: Baseline to week 12. For Phase 2 analysis: Baseline to week 18.
  Parkinson's Anxiety Scale (PAS) is a 12-item validated observer or patient-rated scale consisting of three subscales for persistent anxiety, episodic anxiety, and avoidance behavior in patients with Parkinson Disease. Participants are asked to rate on a scale of 0 (not or never) and 4 (severe or almost always).

SECONDARY OUTCOMES:
Change in Perceived Stress Scale (PSS) | For Phase 1 analysis: Baseline to 6 weeks. For Phase 2 analysis: Baseline to 18 weeks.
  PSS is a 10-question validated instrument that assesses stress. Participants are asked to rate on a scale of 0 (never) to 4 (very often) how often they agree with various statements.
Change in GRID-Hamilton Depression Scale (HAMD) | For Phase 1 analysis: Baseline to 6 weeks. For Phase 2 analysis: Baseline to 18 weeks.
  The GRID-HAMD-17 is used to measure the frequency and intensity of depressive symptoms. Participants are asked to rate frequency of each statement on a scale from "Absent or clinically insignificant" to "Almost all the time." Rating for intensity is on a scale from Absent to Very Severe.
Change in MDS-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) | For Phase 1 analysis: Baseline to week 12. For Phase 2 analysis: Baseline to week 18.
  This is a four-part survey designed for patients with Parkinson Disease. Part I covers non-motor experiences of daily living, Part II covers motor experiences of daily living, Part III covers motor examination and Part IV covers motor complications.

CONTACTS AND LOCATIONS:
Overall Officials: Balachundar Subramaniam, MD, MPH, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Centre, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rangasamy V, Thampi Susheela A, Mueller A, F H Chang T, Sadhasivam S, Subramaniam B. The effect of a one-time 15-minute guided meditation (Isha Kriya) on stress and mood disturbances among operating room professionals: a prospective interventional pilot study. F1000Res. 2019 Mar 26;8:335. doi: 10.12688/f1000research.18446.1. eCollection 2019. PMID 32665843
- [Background] Rain M, Subramaniam B, Avti P, Mahajan P, Anand A. Can Yogic Breathing Techniques Like Simha Kriya and Isha Kriya Regulate COVID-19-Related Stress? Front Psychol. 2021 Apr 15;12:635816. doi: 10.3389/fpsyg.2021.635816. eCollection 2021. PMID 33935886
- [Background] Schneider RB, Auinger P, Tarolli CG, Iourinets J, Gil Diaz MC, Richard IH. Change in the Parkinson Anxiety Scale correlates with change in other clinical measures of anxiety over time. Clin Park Relat Disord. 2021 Dec 13;6:100126. doi: 10.1016/j.prdoa.2021.100126. eCollection 2022. PMID 34977549